CLINICAL TRIAL: NCT06377085
Title: Repurposing 5-Azacytidine for the Treatment of Muscle Contractures in Children With Cerebral Palsy
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Andrea Domenighetti, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 809325
Record Dates: First submitted 2024-03-05; First posted 2024-04-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy; Contracture
Keywords: 5-Azacytidine; Azacitidine; Contracture; Muscle
MeSH Terms: conditions — Cerebral Palsy; Contracture | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: For this Phase 1 trial, we will conduct a dose-escalation study in children having CP who receive 5-Azacytidine (AZA) via a single subcutaneous (SQ) injection two weeks before their surgery, already scheduled to release their contractures. We will use a "3 + 3" dose-escalation design where decisions are based on the rate of toxicity at the current dose level independently from prior dose levels. The primary goal of this study is to determine a Maximum Tolerated Dose (MTD), which will be the highest dose level at which less or equal of 33% of patients experience Dose-Limiting Toxicity (DLT).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- AZA 10mg/m^2 (Experimental): 5-Azacytidine, subcutaneous injection, 10mg/m^2, one subcutaneous injection for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: 5-Azacytidine 10mg/m^2
- AZA 20mg/m^2 (Experimental): 5-Azacytidine, subcutaneous injection, 20mg/m^2, one subcutaneous injection for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: 5-Azacytidine 20mg/m^2
- AZA 35mg/m^2 (Experimental): 5-Azacytidine, subcutaneous injection, 35mg/m^2, one subcutaneous injection for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: 5-Azacytidine 35mg/m^2
- AZA 75mg/m^2 (Experimental): 5-Azacytidine, subcutaneous injection, 75mg/m^2, one subcutaneous injection for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: 5-Azacytidine 75mg/m^2
- Placebo for 10mg/m^2 (Placebo Comparator): Placebo, subcutaneous injection, 10mg/m^2, one subcutaneous injection without the active treatment for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: Placebo for the AZA 10mg/m^2
- Placebo for 20mg/m^2 (Placebo Comparator): Placebo, subcutaneous injection, 20mg/m^2, one subcutaneous injection without the active treatment for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: Placebo for the AZA 20mg/m^2
- Placebo for 35mg/m^2 (Placebo Comparator): Placebo, subcutaneous injection, 35mg/m^2, one subcutaneous injection without the active treatment for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: Placebo for the AZA 35mg/m^2
- Placebo for 75mg/m^2 (Placebo Comparator): Placebo, subcutaneous injection, 75mg/m^2, one subcutaneous injection without the active treatment for duration of study (estimated at 46 - 76 days)
  Interventions: Drug: Placebo for the AZA 75mg/m^2

INTERVENTIONS:
Drug: Placebo for the AZA 10mg/m^2 — Placebo control group for the 10mg/m^2, one-time subcutaneous injection without the active treatment.
  Arms: Placebo for 10mg/m^2
Drug: Placebo for the AZA 20mg/m^2 — Placebo control group for the 20mg/m^2, one-time subcutaneous injection without the active treatment.
  Arms: Placebo for 20mg/m^2
Drug: Placebo for the AZA 35mg/m^2 — Placebo control group for the 35mg/m^2, one-time subcutaneous injection without the active treatment.
  Arms: Placebo for 35mg/m^2
Drug: Placebo for the AZA 75mg/m^2 — Placebo control group for the 75mg/m^2, one-time subcutaneous injection without the active treatment.
  Arms: Placebo for 75mg/m^2
Drug: 5-Azacytidine 10mg/m^2 — 5-Azacytidine 10mg/m^2, one-time subcutaneous injection
  Arms: AZA 10mg/m^2
Drug: 5-Azacytidine 20mg/m^2 — 5-Azacytidine 20mg/m^2, one-time subcutaneous injection
  Arms: AZA 20mg/m^2
Drug: 5-Azacytidine 35mg/m^2 — 5-Azacytidine 35mg/m^2, one-time subcutaneous injection
  Arms: AZA 35mg/m^2
Drug: 5-Azacytidine 75mg/m^2 — 5-Azacytidine 75mg/m^2, one-time subcutaneous injection
  Arms: AZA 75mg/m^2

SUMMARY:
In this controlled dose-escalation study, we will study the initial safety, biological properties, and potential efficacy of 5-azacytidine (AZA). Our overarching aspiration is for AZA to evolve into an approved pharmacological treatment, fostering muscle growth and enhancing body movement, ultimately contributing to an improved quality of life in children with CP.

The main questions this study aims to answer are:

1. What is the optimal dose of AZA injection that can be used safely in children with CP?
2. Can the optimal safe dose of AZA improve the function of muscle-generating stem cells in children with CP?

Each participant will have up to five research visits over the course of the study duration, in which they will participate in: blood draws, pregnancy test(s) (if applicable), medical assessments, and a muscle biopsy during a surgery for muscle contractures.

Researchers will compare participants with four different dosages of AZA injections to those with four different dosages of placebo injections. A placebo is a look-alike substance that contains no active drug. They will see if a single injection of AZA at a standard concentration currently approved by the FDA to treat myelodysplastic syndromes, can also safely improve muscle growth and function in children with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) has an enduring impact on the development of the muscles after birth. Research showed that a drug that is currently approved by the FDA to treat myelodysplastic syndromes in adults and children, can be potentially adapted ("repurposed") to support muscle growth. In a controlled dose-escalation study, we will study the preliminary safety, biological properties, and efficacy of this drug, called 5-Azacytidine (AZA). Our hope and overarching expectations are that one day AZA will become a new approved pharmacological treatment to support muscle growth and improve body movement and quality of life in children with CP.

Research participants will have five study visits.

1. The first study visit will be a screening within 30 days of the baseline visit and will determine eligibility for the study. The participant will have their blood drawn to check for normal kidney and liver functioning, do a pregnancy test (if applicable), and then the researcher will complete a medical assessment.
2. If the participant is eligible, they will be invited to a second study visit approximately 15 days prior to their scheduled surgery for contracture release. At this visit, the participants will get their blood drawn, do a pregnancy test (if applicable), have a medical assessment performed, and receive their injection. The injection will be a single sub-cutaneous shot in their leg, near the muscle group that will undergo surgical repair.
3. The third visit will be at the participant's scheduled surgery. A small sample of the muscle (i.e., about the size of a pencil eraser) will be surgically removed by the researcher from a muscle group that is already exposed during the procedure. The biopsy will add approximately two to five minutes to the overall procedure time. The participant will also have their blood drawn.
4. The participants will be seen approximately one week after their surgery to complete a medical assessment.
5. The last visit will be about four weeks after the surgery at their post-operative appointment. At this visit, the participant will have their blood drawn and complete a medical assessment to test their range of motion following the surgery.

The amount of blood drawn at each time point will be approximately 3 mL, equating to 12 mL of blood total (less than a tablespoon). The purpose of the blood draws is to evaluate safety and biological efficacy of the study drug. The medical assessment will consist of range of motion assessment and wound check performed by the clinicians. These are the same assessments that the clinicians would typically do as part of usual care prior to and after surgery. The purpose of the medical assessment is to evaluate the efficacy of the study drug and ensure the surgical site is healing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cerebral palsy.
2. Either achilles or hamstring spasticity with contracture necessitation surgical lengthening.
3. Between 2 and 18 years of age
4. Normal renal and liver function as defined by NCI-CTCAE criteria.71

   a. Renal Function (Grade 0 - Normal): i. Creatinine: Within the normal range or ≤ 1.0 times the upper limit of normal (ULN).

   ii. Glomerular filtration rate (GFR): No significant decrease. b. Liver Function (Grade 0 - Normal): i. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT): Within the normal range or ≤ ULN.

   ii. Total bilirubin: Within the normal range or ≤ 1.0 times ULN
5. A negative pregnancy test for females of childbearing potential*.
6. Females of childbearing potential must agree to use contraception consistently from screening to 6 months after their injection. Highly effective methods of contraception are required for females of childbearing potential:

   1. Total abstinence from sexual intercourse.
   2. Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).
   3. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, which may be oral, intravaginal, or transdermal used in accordance with medical direction.
   4. Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injected, or implanted, and used in accordance with medical direction.
7. Males of childbearing potential** must agree to use contraception consistently from screening until 3 months after the injection. Acceptable methods of contraception for males of childbearing potential are:

   1. Total abstinence from sexual intercourse.
   2. Condom with spermicide (cream, spray, foam, gel, suppository, or polymer film).

      * Female of childbearing potential is defined as a female capable of becoming pregnant, which includes patients who have had their first menstrual cycle (menarche).

        * Male of childbearing potential is defined as a subject who has reached spermarche.

Exclusion Criteria:

1. Active infection.
2. Cardiac disease.
3. Allergy to AZA or mannitol.
4. Patient or family who is non-compliant.
5. Received chemotherapy in the preceding three months.
6. Evidence of a hematologic precondition or other malignancy.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT). | Through study completion, an average of 2 years.
  The percentage of patients experiencing DLT at the predefined dose level will be calculated.
  This will determine the Maximum Tolerated Dose (MTD), which will be the highest dose level at which ≤ 33% of patients experience a DLT. DLT is defined as toxic effects, presumably related to AZA, considered unacceptable due to their severity and/or irreversibility, thereby limiting further dose escalation. Thus, the total number of toxicities and the DLT at each step of dose escalation and possible de-escalation will be reported. The scale for the primary endpoint is binary (occurrence of DLT or not). It is measured as a single endpoint, as it is focused on whether or not the predefined dose level causes DLT.
  The currently recommended clinical dose is 75 mg/m2. For the present study, the following AZA concentrations will be evaluated: 10 mg/m2, 20 mg/m2, 35 mg/m2 and 75 mg/m2. For each dose, 3 experimental and 3 placebo subjects will be recruited.

SECONDARY OUTCOMES:
Satellite Cell Fusion Index. | Through study completion, an average of 2 years.
  Resident muscle-forming stem cells, called Satellite Cells, will be isolated from the muscle biopsy obtained from subjects and cultured in vitro. Satellite Cell Fusion Index quantifies the proportion of these stem cells that will fuse to form new muscle fibers in vitro (multinucleated structures called myotubes). It provides a measure of the efficiency of subjects' satellite cells to contribute to muscle growth, repair and regeneration.
DNA methylation quantification in Satellite Cells and Blood Mononucleated Cells. | Through study completion, an average of 2 years.
  Global DNA methylation analysis will be quantified (% tot DNA in ng) using DNA from Satellite Cell cultures and Blood Mononucleated Cells (isolated form blood) using an ELISA-based global DNA methylation kit.
DNA methylation profiling in Satellite Cells. | Through study completion, an average of 2 years.
  Following Satellite Cell isolation, expansion in culture and DNA extractions, qualitative methylation analysis procedures will be conducted using an Infinium Human MethylationEPIC Beadchip array (Illumina Inc., CA), which targets over 850,000 DNA methylation sites at the dinucleotide (CpG) level throughout the entire genome.

OTHER OUTCOMES:
Chromatin immunoprecipitation sequencing (ChIP-seq), and assay for transposase-accessible chromatin sequencing (ATAC-seq) | Through study completion, an average of 2 years.
  ChIP-seq will facilitate the genome-wide profiling of changes in chromatin structure and transcription factor binding events in response to AZA treatment and muscle contracture development. This technique is particularly as it can identify alterations in DNA methylation patterns and histone modifications associated with Satellite Cell dysfunction and impaired muscle regeneration. Furthermore, ATAC-seq will offer a complementary approach to ChIP-seq by providing information on chromatin accessibility, which reflects regulatory elements such as enhancers and promoters involved in gene expression control.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Domenighetti, PhD, Principal Investigator — Shirley Ryan AbilityLab; Patrick Curran, MD, Principal Investigator — Rady Children's Hospital, San Diego; Richard L. Lieber, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rady Children's Hospital - San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No